CLINICAL TRIAL: NCT03876379
Title: Brain Power Spectral Density Under Propofol and Its Association With Cerebral Fragility, an Objective Means to Estimate the Probability of Presenting Burst Suppression
Brief Title: Brain Power Spectral Density Under Propofol
Acronym: PROBRAIN
Status: Completed | Type: Observational
Sponsor: Joaquim MATEO (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); M3DISIM (Other)
Responsible Party: Sponsor-Investigator, Joaquim MATEO, Clinical professor, Hopital Lariboisière
Organization: Hopital Lariboisière (Other)
Other Study IDs: Brain Spectral 2016
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Radiography; Orthopedic Surgery; Interventional
Keywords: Depth of anesthesia; brain fragility; electrographic suppression; postoperative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the operating room, the state of anesthesia is monitored during general anesthesia-induced hypnosis through EEG-based neuro-monitoring. Recent studies suggest that variables extracted from per-operative EEG change as brain ages. Furthermore, aging is itself an independant factor associated to an increased sensitivity to General Anesthesia (GA). Among fragility sign, per-operative Burst Suppression (BS) has been associated to a poor postoperative cognitive trajectory. The main goal of this observational clinical study is to extend the traditional use of per-operative EEG to the detection and prediction of various degrees of brain fragility, depending on the depth of anesthesia (DoA).

DETAILED DESCRIPTION:
Main objective : Extend the traditional use of per-operative EEG to the detection and prediction of various degrees of brain fragility, depending on the depth of anesthesia (DoA).

Indices derived from the EEG signal, Spectral Edge Frequency 95 (SEF95), Patient State Index (PSI) and Bi-spectral Index (BIS) are now widely used in the operating room to monitor the Depth of Anesthesia (DoA). Recent studies suggest that variables extracted from per-operative EEG change as brain ages. A detailed reading of the quantitative EEG (qEEG) under GA has been recently described depending both on the specific drug used and patients' age. For GA induced with Propofol (2,6 di-isopropylphenol), a GABAergic receptor agonist used in Total Intra Venous Anesthesia (TIVA), the EEG signal under frontal derivations exhibits a specific signature characterized by a powerful alpha band. However, the elderly attenuates these EEG characteristics, which might be the results of a change in thalamic-cortical function and decreased neuronal excitability.

The goal of this observational clinical study is to assess the fragility of a patient under GA and based on the EEG SEF13 characteristics, weighted by the amount of Propofol administered.

Measures are based on EEG signal and subfrequency power spectral densities including alpha band as well as the amount of Propofol, each measured for EEG periods where SEF 95 = 8-13Hz.

Experimental design: This is a single-center, interventional, category I prospective study (minimal risks and constraints)

Population concerned : Patients eligible for interventional neuroradiology or orthopedic surgery performed under GA are selected to participate in this prospective, observational, single-center, routine care study. Patients will be included if they received, for a non-urgent scheduled procedure, a Total IntraVenous Administration (TIVA) anesthesia by Propofol according to the Schnider model combined with a morphine derivative. Minor patients, pregnant women and patients who refused to provide informed consent are excluded from the study. Patients with a BMI > 36 kg/m2 for whom the Schnider model is not validated are also excluded. Patient demographics will be collected during the anesthesia consultation. Total IntraVenous Anesthesia (TIVA) and Target Controlled Infusion (TCI) are used for morphine derivative and Propofol, EEG parameters will be collected from frontal electrodes montage (Fp1, Fp2, F7, F8).

Research Proceedings : Measures are based on EEG signal through routine EEG-based neuro-monitoring and subfrequency power spectral densities including alpha band as well as the amount of Propofol, each measured for EEG periods where SEF95 = 8-13Hz. Standard monitoring (Pulse Oxygen Saturation: SpO2, Heart Rate: HR, Systolic, Diastolic and Mean Arterial Blood Pressure: SBP, DBP, MAP, Temperature, End tidal CO2: (EtCO2) and electro-encephalogram monitoring by the Masimo Sedline monitor (SEF 95, PSI and BS) will be recorded.

General anesthesia is then induced in a standardized manner with a morphine followed by intra-venous administration of Propofol. All the measures are obtained non-invasively.

Individual benefit: There is no benefit for the patient

Collective benefit: Aging is associated to change in cerebral activity and it's crucial to distinguishes fragile patients from normal ones. The tailoring of doses according to the degree of "cerebral fragility" could predict poor postoperative cognitive or behavioral evolution.

Risks and minimal constraints added by the research: No added risk. The procedure is performed according to the usual protocol including routine EEG-based neuro-monitoring All the measures are obtained non-invasively.

For all patients whatever the comorbidities, anesthesia induction will be performed using a target-controlled infusion (Orchestra® Base Primea - Fresenius Kabi France). According to our standard of care, intra-operative episodes of hypotension (mean arterial pressure (MAP) < 65 mmHg or < 80% baseline) are treated by Norepinephrine bolus of 10 μg. For all patients, data from EEG-neuromonitoring and hemodynamic data are collected at the end of the procedure.

Number of selected subjects Selection of patients up to 60 analysable patients Number of Centre : 1 Research Agenda inclusion period: 12 months duration of participation (treatment + follow-up): duration of the interventional neuroradiology or orthopedic procedure: 1 day total duration: 12 months Number of planned inclusions by centre and month : 5 Number of subjects required : 60

Statistics The significance level used in this study chose as 0.05. The values is expressed in percentage for qualitative variables and median (InterQuartile Range: [IQR]) for quantitative variables. All parameters will be recorded and the brain total power spectral density (PT), alpha band power spectral density (Pα) and the Propofol TCI (µg/ml) will be calculated on the entire population. The median value of Pα,PT,PropofolTCI combination will be compared using non-parametric Kruskal Wallis and Man Whitney tests for quantitative data, while qualitative variable will be analyzed based on the Fisher's test. Research on the correlation between age and brain total power spectral is carried out by Pearson's test.

Then analysis will be also performed according to the occurrence of BS during induction of anesthesia. ROC curves will be constructed from univariate logistic régressions. For each univariate regression investigators provided Odd Ratios (OR) given with a 95% Confidence Interval (CI) and Areas Under the Curve (AUC). Multivariate analysis is finally performed with a logistic regression model where explanatory variables are chosen according to the results of the univariate analysis (p-value≤0.1).

The sample size calculation is based on the following assumptions : Assuming an incidence of 40% BS, with a power at 80% and an alpha risk at 5%, it is necessary to include 60 patients to highlight an area under the ROC curve of 80% with a confidence interval width of 0.1.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years scheduled an elective interventional neuroradiology procedure or orthopedic surgery performed under general anesthesia.
* oral agreement obtained from each patient before anesthesia

Exclusion Criteria:

* age <18 years
* an emergency procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years scheduled an elective interventional neuroradiology procedure or orthopedic surgery performed under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-01-24 (Actual); Primary Completion 2016-01-05 (Actual); Study Completion 2016-01-05 (Actual)

PRIMARY OUTCOMES:
Values of Patient State Index (PSI-) are collected from frontal electrodes montage (Fp1, Fp2, F7, F8) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)]]
  For all patients values of Patient State Index (PSI -) will be collected during Total Anesthesia Period (induction and hypnotic periods)
Propofol doses administered with Target Controlled Infusion (TCI in µg/ml) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)]]
  For all patients values of Target Controlled Infusion (TCI in µg/ml ) will be collected during Total Anesthesia Period (induction and hypnotic periods)
Values of Burst Suppression (in % of time) are collected from frontal electrodes montage (Fp1, Fp2, F7, F8) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)]]
  For all patients values of Burst Suppression (in % of time) will be collected during Total Anesthesia Period (induction and hypnotic periods)
Values of the Spectral Edge Frequency (SEF 95 in uV2/Hz) are collected from frontal electrodes montage (Fp1, Fp2, F7, F8) | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)]]
  For all patients values of the Spectral Edge Frequency (SEF 95 in uV2/Hz) will be collected during Total Anesthesia Period (induction and hypnotic periods)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Principal Investigator — HLariboisiere LeTemple